CLINICAL TRIAL: NCT00517023
Title: Eastbourne Syncope Assessment Study II
Acronym: EaSyAS II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastbourne General Hospital (Other)
Collaborators: Transoma Medical (Industry); East Sussex National Health Service Trust, United Kingdom (Unknown)
Responsible Party: Dr AN Sulke, Cardiac Department, Eastbourne General Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 07/Q1907/13; T07-015
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Syncope
Keywords: Implantable Loop Recorder; Home monitoring; Syncope/ Falls Clinic
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ILR + Syncope Clinic (Active Comparator): Patients will have ILR implanted and follow-up in Syncope Clinic
  Interventions: Device: Sleuth Implantable Loop Recorder
- ILR Only (Active Comparator): Patients will have ILR implanted and routine follow up.
  Interventions: Device: Sleuth Implantable Loop Recorder
- Routine Mx + Syncope Clinic (Active Comparator): Patients will receive routine care and management plus follow up in Syncope Clinic
  Interventions: Other: Other
- Routine Mx (Active Comparator): Patients will receive routine care and management
  Interventions: Other: Other

INTERVENTIONS:
Device: Sleuth Implantable Loop Recorder — ILR insertion under aseptic conditions in left pectoral region (local anaesthetic procedure only)
  Arms: ILR + Syncope Clinic; ILR Only
Other: Other — Routine care and tests usually offered for syncope patients.
  Arms: Routine Mx; Routine Mx + Syncope Clinic

SUMMARY:
Syncope (commonly called collapses or blackouts) is defined as loss of consciousness which is transient, self limiting and usually leads to falling.

While the causes of syncope encompass a wide variety of factors, those due to heart rhythm abnormalities are acknowledged to be significantly more serious compared with other causes.

The main aim of the study is to see if it is possible to find the cause of a patient's syncope faster using a device called an implantable loop recorder (ILR), which is implanted under the skin, versus conventional management. The device is slightly larger than a 50 pence coin and records the rhythm of the heart continuously.

Although ILRs are being used widely today, we want to use a new model that is able to relay information to the doctor via wireless technology and internet.

We also want to use ILRs earlier in diagnosing syncope, thereby avoiding unnecessary and lengthy hospital admissions and lowering cost.

Primary aim: To see how soon the ILR detects abnormal heart rhythms or normal ones (in study subjects who faint/ suffer syncope).

Secondary aims are:

1. To see how soon treatment is started once the abnormal rhythm is detected by the ILR.
2. To see which group (patients with ILRs or those receiving conventional tests) receives treatment sooner.
3. To see which group has less subsequent collapses i.e has benefited from appropriate treatment sooner.
4. To assess the cost effectiveness of using the implantable loop recorder more as a diagnostic tool for syncope versus conventional management (it should save many hospital admissions).

DETAILED DESCRIPTION:
The original EaSyAS study (1998) evaluated the use of implantable loop recorders (ILRs) in the diagnosis and management of syncope.This demonstrated a significant increase in successful diagnosis following use of implantable loop recorders. Here there were 442 syncope admissions to Eastbourne in 2001. Diagnostic rate was 42%. In addition, time to diagnosis was quicker and therefore so was introduction of therapy. This resulted in significant increase in time to recurrent syncopal episodes and improved general wellbeing in an unselected population with syncope of an unknown cause.

The "Post-EaSyAS" study evaluated extended (2.5 years) follow up of these patients. The "Tis-EaSyAS" study evaluated 3 different tilt protocols with long term ILR follow up describing the positive predictive value of tilt testing in unexplained syncope.

The EaSyAS II study elaborates further the above by using the ILR to avoid hospital admission and optimise the use of a falls/syncope clinic, potentially improving cost effective diagnosis and management of syncope.

ILRs will be implanted without patient admission and with follow up in a syncope/falls assessment clinic, compared to optimal protocol driven current management.

The ILR used has capabilities to record and transmit heart rhythm abnormalities to a wireless receiver which will then relay the information to the clinician via the internet. It is hoped that this will shorten diagnosis times and speed up commencement of treatment for patients, and will avoid expensive tests and more expensive hospital admissions.

ELIGIBILITY:
Inclusion Criteria:

* Age > = 16 yrs
* Acute syncope presentation to MAU or A+E
* 2 or more unexplained syncopes within the past 24 months including index episode
* Normal baseline ECG
* Absence of co - existing pathology requiring admission

Exclusion Criteria:

* Suspected or known heart disease
* ECG abnormalities suspected of arrhythmic syncope listed in Table 1
* Syncope occurring during exercise
* Syncope causing severe injury
* Family history of sudden death
* Sudden onset palpitations prior to syncope

Table 1: ECG Abnormalities:

* Bifascicular block (defined as LBBB or RBBB combined with left anterior or left posterior fascicular block)
* Other intraventricular abnormalities (QRS duration >= 0.12s)
* Mobitz 1 second degree AV block (Wenckebach)
* Asymptomatic sinus bradycardia (<50 bpm), SA node or sinus pause >= 3s in the absence of negatively chronotropic medications
* Pre-excited QRS with short PR interval (WPW)
* Significantly Prolonged QT interval
* RBBB pattern with ST elevation in V1 - V3 (Brugada Syndrome)
* Negative T waves with ST segment elevation in right precordial leads suggestive of arrythmogenic right ventricular dysplasia
* Significant Q waves (>= 0.02s) suggestive of MI

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-07 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome 1. Time to ECG (objective) diagnosis of syncope | 1 Year

SECONDARY OUTCOMES:
1. Time to ECG directed therapy. 2. Time to introduction of empiric therapy. 3. Time to first post induction syncope. 4. Cost effectiveness analysis. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: A N Sulke, DM FRCP FESC FACC, Principal Investigator — Eastbourne General Hospital
Locations (1):
- Cardiology Department, Eastbourne General Hospital, Eastbourne, East Sussex, United Kingdom